CLINICAL TRIAL: NCT03471351
Title: An Open Label, Phase I/II Study to Evaluate the Safety and Efficacy of RP6530, a Novel PI3K δ/γ Dual Inhibitor Given in Combination With an Anti-PD-1 Therapy, Pembrolizumab in Adult Patients With Relapsed or Refractory cHL
Brief Title: Safety and Efficacy Study of Tenalisib (RP6530) in Combination With Pembrolizumab in Relapsed or Refractory cHL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: At this point, the current study in HL does not fit into clinical development and regulatory strategy.
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530+Pembrolizumab-1701
Record Dates: First submitted 2018-02-15; First posted 2018-03-20 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; RP6530; Pembrolizumab; Tenalisib
MeSH Terms: conditions — Hodgkin Disease | interventions — tenalisib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenalisib+Pembrolizumab (Experimental): Participants receive Tenalisib in escalating doses Orally BID and pembrolizumab as a fixed dose intravenously (IV) in Escalation and Expansion.
  Interventions: Drug: Tenalisib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Tenalisib — Tenalisib, BID, orally and Pembrolizumab 200 mg IV Q3W
  Other Names: RP6530
Biological: Pembrolizumab — Tenalisib, BID, orally and Pembrolizumab 200 mg IV Q3W

SUMMARY:
To characterize safety, tolerability and to establish the maximum tolerated dose (MTD) for Tenalisib in combination with Pembrolizumab in patients with cHL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years on the day of signing informed consent.
2. Histologically confirmed diagnosis of cHL.
3. Disease status as defined as.

   * Refractory patients who are naïve to anti-PD-1/PDL-1 therapy OR Relapsed after 3 or more lines of therapies; and are naïve to anti-PD-1/PDL-1 therapy OR
   * Patients currently on Pembrolizumab and achieve a less than complete response
4. Must have ECOG performance status of 0 or 1
5. At least one bi-dimensional measurable lesion with minimum measurement of > 15 mm in the longest diameter.
6. Toxicities related to prior therapy must have returned to Grade 1 or less, except for alopecia.

   1. Adequate bone marrows, liver and renal function as assessed by the following laboratory requirements. Hemoglobin ≥8.0 g/dL (may not be transfused or treated with erythropoietin in preceding week to maintain or exceed this level)
   2. Absolute neutrophil count (ANC) ≥1,000/µL
   3. Platelet count ≥75,000/μL
   4. Total bilirubin ≤1.5 times the ULN (or ≤3 x ULN, if patient has Gilbert syndrome)
   5. ALT and AST ≤2.5 x ULN
   6. Serum creatinine ≤ 1.5 x ULN or CrCl > 60 ml/min (Cockcroft-Gault formula)
7. Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential
8. Provide written informed consent prior to any study-specific screening procedures.
9. Willingness and capability to comply with the requirements of the study.

Exclusion Criteria:

1. Patient receiving anticancer therapy (e.g. chemotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization) ≤3 weeks or 5 half-lives (whichever is shorter) prior to C1D1,
2. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
3. Radiotherapy within the last 21 days prior to C1D1 (limited field palliative radiation is allowed if ≥ 14 days prior to C1D1);
4. Investigational drug therapy outside of this trial during or within 3 weeks prior to C1D1.
5. Patients with Allo-SCT on active GVHD or immunosuppression therapy within 3 months prior to C1D1.
6. Patient with active autoimmune disease or any medical condition requiring the use of systemic immunosuppressive medications .
7. Pregnancy or lactation.
8. Known clinically active CNS involvement.
9. Evidence of active Hepatitis B, active Hepatitis C infection (HCV) or cytomegalovirus (CMV) or known history of HIV.
10. Subjects with concomitant second malignancies
11. Patient with any active immune toxicity of Grade 1 or greater or any other severe or Grade 3 treatment-related adverse event.
12. History of Grade 4 anaphylactic reaction to monoclonal antibody therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for Tenalisib in combination with Pembrolizumab in patients with cHL | 21 days
  The MTD was defined as the highest dose level at which no more than 1 in 6 participants experienced a dose-limiting toxicity (DLT) during the first 21-day cycle of treatment.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 21 days
  Assessment of Cmax in subjects treated with RP6530 and pembrolizumab combination
Overall response rate (ORR) with Tenalisib and Pembrolizumab combination | 12 weeks
  No of patients with partial and complete response
Duration of Response (DoR) with Tenalisib and Pembrolizumab combination | 12 weeks
  The time period from the response achieved in patient until the disease progression.
Progression free survival (PFS) with Tenalisib and Pembrolizumab combination | 12 weeks
  Progression-free survival was defined as the time from enrollment in the study to disease progression
Conversion Rate with Tenalisib and Pembrolizumab combination | 12 weeks
  Defined as improved outcome status (i.e Improve from PR to CR or from SD to PR)
Proportion of patients achieving CR and PR with Tenalisib and Pembrolizumab combination | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Rhizen Pharmaceuticals investigational trial site; Karmanos Cancer Institute,, Detroit, Michigan
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No